CLINICAL TRIAL: NCT07064330
Title: Next Generation Flow Cytometry for Global Immunological Profile, Response And Toxicity Biomarker Signatures in Cutaneous Squamous Cell Carcinoma Under CEmiplimab Treatment.
Brief Title: Next-gen Flow Cytometry to Find Immune Profiles, Treatment Response, and Toxicity Markers in Skin Cancer Patients Treated With Cemiplimab.
Acronym: NGF-GRACE
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Carlos III Health Institute (Other Government); University of Salamanca (Other)
Responsible Party: Sponsor
Other Study IDs: NGF-GRACE Study; E.O. 24/841 (Other: Ethics Committee for Clinical Research of the Health Area of Salamanca (CEIm))
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cutaneous Squamous Cell Carcinoma (CSCC)
Keywords: Cemiplimab; Rhapsody Single Cell System; Tumor Microenvironment
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Whole perypheral blood and tumor samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: All enrolled patients will receive cemiplimab as part of standard clinical care for advanced cutaneous squamous cell carcinoma (CSCC). Cemiplimab is not assigned by the study but is administered as per physician's decision in routine practice.
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — 350 mg IV every 3 weeks as per standard of care. Patients are observed prospectively for biomarkers of response and toxicity during cemiplimab treatment.

SUMMARY:
Cutaneous squamous cell carcinoma (CSCC) is the second most frequent cancer in humans, it exhibits a high tumor mutational burden and is more common in immunocompromised patients, which aimed to explore the impact of immunotherapy in this cancer. CSCC shows good response to anti-PD1 immunotherapy, and cemiplimab is the first FDA-approved and the only EMA-approved treatment for this tumor. However, 50% of patients won't respond to anti-PD1 and to date there is little evidence on the reasons for such a lack of effectiveness. Also, anti-PD1 immunotherapy is very safe, but some patients will develop adverse events, and anticipating severe adverse events might help in patients' management. The NGF-GRACE project aims to find biomarkers of response and toxicity, both in the blood and the tumor, using advanced technologies. The goal is to move towards more personalized treatments, better select patients, predict side effects, and improve our understanding of the immune system in CSCC.

DETAILED DESCRIPTION:
The NGF-GRACE project focuses on identifying biomarkers of response and toxicity in patients with advanced cutaneous squamous cell carcinoma (CSCC) undergoing anti-PD1 treatment, being cemiplimab the unique approved drug in Europe. CSCC, characterized by a high mutational burden and increased risk in immunosuppressed patients, has exhibited significant sensitivity to anti-PD1 immunotherapy. By employing cutting-edge technologies such as Next Generation Flow Cytometry and the BD Rhapsody Single Cell System, the study aims to assess the immunological profile in peripheral blood and in the tumor tissue. The ultimate goal is to advance towards a more individualized therapeutic approach, identifying biomarkers that enhance patient selection, anticipate adverse events, and address knowledge gaps in the CSCC tumor immunology.

Background and Rationale CSCC is a type of skin cancer with one of the highest mutational burdens among solid tumors, making it particularly sensitive to immunotherapy, especially PD-1 blockade. Cemiplimab, an anti-PD-1 antibody, has become the first FDA and EMA-approved treatment for advanced CSCC. However, response rates are variable, with around 50% of patients showing clinical benefit. There is an urgent need to identify predictive biomarkers to guide patient selection, anticipate toxicity, and understand resistance mechanisms.

Study Objectives The main objective is to identify biomarker of response and toxicity to cemiplimab in patients with advanced cutaneous squamous cell carcinoma

Study Design The study will enroll approximately 30 patients with locally advanced or metastatic CSCC who will start cemiplimab treatment. Peripheral blood and tumor samples will be collected. A preliminary phase with 5 patients will define optimal sampling timepoints.

Methods Peripheral blood will be analyzed using Next Generation Flow Cytometry (NGF), applying a custom-designed 40-color antibody panel to characterize innate and adaptive immune cells. Also, soluble biomarkers will be evaluated. Single-cell technologies will be implemented for tumor evaluation.

Endpoints and Data Analysis Clinical response will be measured using RECIST 1.1, and toxicity will follow CTCAE v5.0. Statistical analyses will correlate immune profiles with outcomes using appropriate tests (e.g., chi-square, t-tests, ANOVA, Kaplan-Meier survival analysis).

Ethical Considerations The study complies with the Declaration of Helsinki, GCP, and GDPR. Informed consent is mandatory, and data confidentiality is ensured. Samples and data will only be used for approved research purposes.

Impact The NGF-GRACE project seeks to advance precision immunotherapy in CSCC by identifying predictive biomarkers that can improve patient selection, predict adverse events, and inform new therapeutic strategies. The study's innovative technologies and comprehensive design position it to fill critical knowledge gaps in CSCC immuno-oncology.

ELIGIBILITY:
- Inclusion criteria At least 18 years old

Hepatic function:

1. Total bilirubin ≤1.5x upper limit of normal (ULN) (or ≤3x ULN, if liver metastases).
2. Patients with Gilbert's Disease and total bilirubin up to 3x ULN may be eligible after communication with and approval from the medical monitor
3. Transaminases ≤3x ULN (or ≤5x ULN, if liver metastases)
4. Alkaline phosphatase (ALP) ≤2.5x ULN (or ≤5x ULN, if liver or bone metastases) Renal function: Serum creatinine ≤2x ULN or estimated creatinine clearance >35 mL/min (according the method of Cockcroft and Gault) Creatine phosphokinase (CPK) (also known as CK [creatine kinase]) elevation ≤ grade 2

Bone marrow function:

a. Hemoglobin ≥9.0 g/dL b. Absolute neutrophil count (ANC) ≥1.5 x 109/L c. Platelet count ≥75 x 109/L Anticipated life expectancy >12 weeks

- Exclusion criteria:

1. - Patient who refuses to participate in the study.
2. Being unsuitable for cemiplimab treatment
3. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events (irAEs). The following are not exclusionary: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism requiring only hormone replacement, or psoriasis that does not require systemic treatment.
4. Untreated brain metastasis(es) that may be considered active.

   a. Note in clarification: Patients with previously treated brain metastases may participate provided that the lesion(s) is (are) stable (without evidence of progression for at least 6 weeks on imaging obtained in the screening period), and there is no evidence of new or enlarging brain metastases, and the patients do not require any immunosuppressive doses of systemic corticosteroids for management of brain metastasis(es) within 28 days of the first dose of REGN2810cemiplimab.
5. Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of REGN2810cemiplimab

   a. Note in clarification: Patients who require brief courses of steroids (eg, as prophylaxis for imaging studies due to hypersensitivity to contrast agents) are not excluded
6. Active infection requiring therapy, including positive tests for human immunodeficiency virus (HIV)-1 or HIV-2 serum antibody, hepatitis B virus (HBV), or hepatitis C virus (HCV)
7. History of pneumonitis within the last 5 years
8. Any anticancer treatment other than radiation therapy (chemotherapy, targeted systemic therapy, imiquimod, photodynamic therapy), investigational or standard of care, within 30 days of the initial administration of REGN2810 cemiplimab or planned to occur during the study period
9. History of documented allergic reactions or acute hypersensitivity reaction attributed to antibody treatments
10. Patients with allergy or hypersensitivity to REGN2810 cemiplimab or to any of the excipients must be excluded.
11. Patients with a history of solid organ transplant (patients with prior corneal transplants may be allowed to enroll after discussion with and approval from the medical monitor)
12. Breastfeeding
13. Positive serum pregnancy test (a false positive pregnancy test, if demonstrated by serial measurements and negative ultrasound, will not be exclusionary, upon communication with and approval from the medical monitor)
14. Receipt of live vaccines (including attenuated) within 30 days of first study treatment
15. Women of childbearing potential (WOCBP)*, or sexually active men, who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment prior to the start of the first treatment, during the study, and for at least 6 months after the last dose.

    Optional criteria, depending on the therapy being investigated:
16. Prior treatment with an agent that blocks the PD-1/PD-L1 pathway (If a study is addressing prior unsuccessful treatment with PD-1/PD-L1 inhibitor, it is suggested to exclude patients who had suffered from ≥grade 3 irAE during previous treatment)
17. Prior treatment with other systemic immune-modulating agents within fewer than 28 days prior to the first dose of REGN2810cemiplimab. Examples of immune-modulating agents include therapeutic vaccines, cytokine treatments, or agents that target cytotoxic T-lymphocyte antigen 4 (CTLA-4), 4-1BB (CD137), or OX-40.

    1. Note in clarification: Prior treatment with imiquimod or other topical or intralesional immune modulators will not be exclusionary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient who is going to be treated with cemiplimab is a potential candidate for this study considering the inclusion and exclusion criteria of the registry study, included in SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Biomarker signature associated with cemiplimab response | Up to 6 months from treatment initiation
  Identification of peripheral blood and tumor immune biomarkers (cellular and soluble) that correlate with objective response to cemiplimab. Immune biomarkers to be reported include:
  1. Peripheral blood biomarkers (cellular and soluble):
     * Cellular biomarkers include: CD4⁺, CD8⁺ and T cells, B and plasma cells, NK cells, monocytes, dendritic cells and other myeloid populations, functional and checkpoint markers (e.g. PD-1, HLA-DR).
     * Soluble biomarkers (cytokines and chemokines): IL-2, IL-6, IL-10, IFN-γ, TNF-α, Chemokines (CXCL9, CXCL10, CCL2, and CCL5).
  2. Tumor tissue biomarkers (single-cell multi-omics):
     * Cellular biomarkers: CD3, CD4, CD8, CD11c, CD14, CD16, CD19, CD25, CD27, CD28, CD45RA, CD56, CD62L, CD127, CD134, CD137, CD161, CD183, CD185, CD186, CD196, CD197, CD272, CD278, CD279, CD357, CD366, HLA-DR, IgD and IdM.
     * Transcriptomic biomarkers:
  Single-cell transcriptome data (WTA library) will be generated to explore gene expression profiles associated with immune response.
Best Overall Response (BOR) | From baseline to end of treatment (up to 12 months)
  Proportion of patients with complete response (CR) or partial response (PR) according to RECIST v1.1 criteria, as assessed during cemiplimab treatment.
Immune-related toxicity rate | From first infusion until 90 days after last dose of cemiplimab
  Descripción: Incidence and severity of immune-related adverse events (irAEs) according to CTCAE v5.0, and their association with baseline immune profiles.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 18 months
  Time from cemiplimab initiation to disease progression or death from any cause.
Overall Survival (OS) | Up to 24 months
  Time from cemiplimab initiation to death from any cause.
Analysis of transcriptomic and proteomic immune profiling of tumor-infiltrating cells | From pre-treatment biopsy to post-infusion sample (up to 3 months)
  Single-cell analysis of tumor samples before and during treatment, identifying profiles associated with response or resistance.
Correlation between tumor and blood immune biomarkers | Up to 6 months
  Association between immune signatures in peripheral blood and those found in the tumor microenvironment. Immune biomarkers to be reported include: 1. Peripheral blood biomarkers (cellular and soluble): - Cellular biomarkers include: CD4⁺, CD8⁺ and T cells, B and plasma cells, NK cells, monocytes, dendritic cells and other myeloid populations, functional and checkpoint markers (e.g. PD-1, HLA-DR). - Soluble biomarkers (cytokines and chemokines): IL-2, IL-6, IL-10, IFN-γ, TNF-α, Chemokines (CXCL9, CXCL10, CCL2, and CCL5). 2. Tumor tissue biomarkers (single-cell multi-omics): - Cellular biomarkers: CD3, CD4, CD8, CD11c, CD14, CD16, CD19, CD25, CD27, CD28, CD45RA, CD56, CD62L, CD127, CD134, CD137, CD161, CD183, CD185, CD186, CD196, CD197, CD272, CD278, CD279, CD357, CD366, HLA-DR, IgD and IdM. - Transcriptomic biomarkers: Single-cell transcriptome data (WTA library) will be generated to explore gene expression profiles associated with immune response.
Treatment discontinuation due to toxicity | From first dose to end of treatment (up to 12 months)
  Rate and reasons for cemiplimab discontinuation related to adverse events.

OTHER OUTCOMES:
Change in immune cell subpopulations over time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Longitudinal changes in peripheral immune cell subpopulations measured by spectral flow cytometry (NGF).
Change in soluble immune markers over time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Longitudinal variation of cytokines and chemokines in serum analyzed by Luminex.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cañueto, Medical Degree in Dermatology, Principal Investigator — Centro Asistencial Universitario de Salamanca (CAUSA)
Locations (1):
- Complejo Asistencial Universitario de Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in future publications (after de-identification) will be made available upon reasonable request. This includes data related to baseline characteristics, treatment administration, toxicity, tumor response, survival outcomes, and quality of life assessments
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available starting 12 months after publication of primary results and for a minimum of 5 years thereafter.
Access Criteria: Sharing Access Criteria: Qualified researchers with a methodologically sound proposal, as determined by the study steering committee, will be able to access the data. Requests should be directed to the study PI. A data access agreement will be required.